CLINICAL TRIAL: NCT05366751
Title: An Open-label Study of the Long-term Safety and Tolerability of SAGE-324 in Participants With Essential Tremor
Brief Title: A Study to Evaluate the Long-term Safety and Tolerability of SAGE-324 in Participants With Essential Tremor
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Internal company decision
Sponsor: Sage Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 324-ETD-303
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Results first posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Essential Tremor
Keywords: SAGE-324
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SAGE-324 60 mg (Experimental): Participants will receive SAGE-324 15 milligrams (mg) from Day 1 to Day 14, followed by up-titration to 30 mg from Day 15 to Day 28, then to 45 mg from Day 29 to Day 42, and then 60 mg starting on Day 43, orally, once daily.
  Interventions: Drug: SAGE-324

INTERVENTIONS:
Drug: SAGE-324 — SAGE-324 oral tablets

SUMMARY:
The primary purpose of this study is to evaluate the long-term safety and tolerability of SAGE-324 in participants with essential tremor (ET).

ELIGIBILITY:
Inclusion Criteria:

1. Participant is in good physical health and has no clinically significant findings (excluding ET) that may impact their ability to participate in the study, as determined by the investigator, on physical examination, 12-lead electrocardiogram (ECG), or clinical laboratory tests.
2. Participant has a clinician-confirmed diagnosis of ET in compliance with all the following criteria:

   1. Duration of at least 3 years
   2. Absence of other neurological signs, such as dystonia, ataxia, parkinsonism, task- and position-specific tremors, sudden tremor onset, or evidence of stepwise deterioration of tremor
   3. Absence of historical or clinical evidence of tremor with psychogenic origin (including, but not limited to, eating disorders and major depression)
3. Participant has completed the planned end of treatment (EOT) visit and was not early terminated during the planned Treatment Period in another SAGE-324 study.
4. Participant is willing to limit use of alcohol to 2 units per day for males and 1 unit per day for females starting at least 1 week prior to Day 1 and through the End of Study (EOS) Visit.

   1. Participant will limit alcohol use to at least 2 hours before self-administration of investigational product (IP) in the evening.
   2. Participant will not use alcohol starting 24 hours prior to scheduled in-clinic study visits until all assessments have been completed.
5. Participant is willing to maintain prestudy consumption of products that contain nicotine starting at least 1 week prior to Day 1 and through EOS Visit.

Exclusion Criteria:

1. Participant has presence of alcohol withdrawal state.
2. Participant has had direct or indirect injury or trauma to the nervous system within 3 months before the onset of tremor.
3. Participant is taking and unable to discontinue the use of primidone at least 7 days prior to administration of the first dose of SAGE-324.
4. Participant has a history (within 3 years of Screening) or ongoing oncologic disease, excluding skin cancers (squamous or basal cell carcinoma) for which treatment has been completed and any carcinoma in situ.
5. Participant has an ongoing clinically relevant medical or psychiatric condition that, in the judgment of the investigator, is not well managed and poses a risk for participation in the study.
6. Participant has history of substance dependence and/or abuse prior to Screening, has a positive screen for drugs of abuse at Screening or predose on Day 1. Participants with nicotine use disorder that impacts their tremor are excluded.
7. Participant has a known allergy to SAGE-324 or any excipient.
8. Female participant has a positive pregnancy test or confirmed pregnancy or is breastfeeding.
9. Participant has had exposure to another investigational drug or device within 30 days or 5 half-lives of the other investigational drug, whichever is longer, prior to the Day 1 visit and for the duration of the study.
10. Participant has a history of suicidal behavior within 2 years or answers "YES" to questions 3, 4, or 5 on the C-SSRS at Screening or at Day 1 or is currently at risk of suicide in the opinion of the investigator.
11. Participant has any condition or comorbidity that in the opinion of the investigator would limit or interfere with the participant's ability to complete or partake in the study.
12. Participant has used any known moderate or strong cytochrome P450 3A4 inhibitors and/or inducers within 14 days or 5 half-lives (whichever is longer) prior to Day 1 or consumed grapefruit juice, grapefruit, Seville oranges, or St. John's Wort or products containing these within 30 days prior to Day 1 and is unwilling to refrain from taking these medications or foods for the duration of dosing. Use of mild cytochrome inhibitors and/or inducers may be permitted.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Sage Investigational Site, Hoover, Alabama
  - Sage Investigational Site, Scottsdale, Arizona
  - Sage Investigational Site, Fountain Valley, California
  - Sage Investigational Site, Fullerton, California
  - Sage Investigational Site, Los Angeles, California
  - Sage Investigational Site, Englewood, Colorado
  - Sage Investigational Site, Boca Raton, Florida
  - Sage Investigational Site, Bradenton, Florida
  - Sage Investigational Site, Coral Springs, Florida
  - Sage Investigational Site, Hollywood, Florida
  - Sage Investigational Site, Miami, Florida
  - Sage Investigational Site, Naples, Florida
  - Sage Investigational Site, Orlando, Florida
  - Sage Investigational Site, Tampa, Florida
  - Sage Investigational Site, Atlanta, Georgia
  - Sage Investigational Site, Decatur, Georgia
  - Sage Investigational Site, Kansas City, Kansas
  - Sage Investigational Site, Lexington, Kentucky
  - Sage Investigational Site, Shreveport, Louisiana
  - Sage Investigational Site, Boston, Massachusetts
  - Sage Investigational Site, Farmington Hills, Michigan
  - Sage Investigational Site, New York, New York
  - Sage Investigational Site, Asheville, North Carolina
  - Sage Investigational Site, Cincinnati, Ohio
  - Sage Investigational Site, Dayton, Ohio
  - Sage Investigational Site, Tulsa, Oklahoma
  - Sage Investigational Site, Memphis, Tennessee
  - Sage Investigational Site, Austin, Texas
  - Sage Investigational Site, Fort Worth, Texas
  - Sage Investigational Site, Houston, Texas
  - Sage Investigational Site, Katy, Texas
  - Sage Investigational Site, Round Rock, Texas
  - Sage Investigational Site, West Falls Church, Virginia
  - Sage Investigational Site, Kirkland, Washington
  - Sage Investigational Site, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 29 investigative sites in the United States from 03 June 2022 to 10 September 2024.
Pre-assignment Details: This was a single-arm study and all participants received SAGE-324 according to a predefined up-titration scheme as follows: 15 milligrams (mg) from Day 1 to Day 14, followed by up-titration to 30 mg from Day 15 to Day 28, then to 45 mg from Day 29 to Day 42, and then 60 mg starting on Day 43. Data were collected and reported in single arm for each participant who started treatment as specified and either completed or discontinued study.
Groups:
- SAGE-324: Participants received SAGE-324 15 mg from Day 1 to Day 14, followed by up-titration to 30 mg from Day 15 to Day 28, then to 45 mg from Day 29 to Day 42, and then 60 mg starting on Day 43, orally, once daily.
Period: Overall Study
Arm/Group | SAGE-324
Started | 97
Completed | 0
Not Completed | 97
Not completed — Adverse Event | 25
Not completed — Physician Decision | 3
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 14
Not completed — Study Terminated by Sponsor | 50
Not completed — Site Terminated by Sponsor | 3

BASELINE CHARACTERISTICS:
Population: The Safety Set included all participants who were administered at least one dose of SAGE-324.
Arm/Group | SAGE-324
Number analyzed (Participants) | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (10.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 91
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 90
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a medicinal (investigational) product whether or not related to the medicinal (investigational) product. A TEAE is defined as an AE with onset after the first dose of IP, or any worsening of a pre-existing medical condition/AE with onset after the start of IP and throughout the study.
Time Frame: Up to 814 days
Population: The Safety Set included all participants who were administered at least one dose of SAGE-324. All participants received SAGE-324 according to a predefined up-titration scheme. Data was collected and reported in single arm for each participant who started treatment as specified and either completed or discontinued study.
Measure: Count of Participants; unit: Participants
Arm/Group | SAGE-324
Number analyzed (Participants) | 97
Participants | 86

2. Secondary Outcome: Number of Participants With Potentially Clinically Significant (PCS) Vital Sign Measurements: Heart Rate, Systolic Blood Pressure (SBP), and Diastolic Blood Pressure (DBP)
Description: Number of participants with PCS postbaseline vital sign values are summarized for categories: supine and standing (1 and 3 minutes [min]) heart rate - maximum absolute value greater than (>)120 beats/min, minimum absolute value less than (<)40 beats/min. Supine and standing (1 and 3 min) SBP - maximum absolute value >180 millimeters of mercury (mmHg), minimum absolute value <90 mmHg, and increase or decrease from baseline of greater than or equal to (≥)30 mmHg; supine and standing (1 and 3 min) DBP - maximum absolute value >110 mmHg, minimum absolute value <50 mmHg, and increase or decrease from baseline of ≥20 mmHg. Only those categories where at least 1 participant met the PCS criterion at least once during postbaseline duration are reported.
Time Frame: Up to 814 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SAGE-324
Number analyzed (Participants) | 97
Participants
  Heart Rate, Supine, >120 beats/min | 1
  Heart Rate, Standing 1 min, >120 beats/min | 2
  Heart Rate, Standing 3 min, <40 beats/min | 1
  Heart Rate, Standing 3 min, >120 beats/min | 1
  SBP, Supine, Change From Baseline (CFB) ≥30 mmHg | 7
  SBP, Supine, CFB less than or equal to (≤ -30) mmHg | 6
  SBP, Standing 1 min, <90 mmHg | 5
  SBP, Standing 1 min, CFB ≥30 mmHg | 6
  SBP, Standing 1 min, CFB ≤ -30 mmHg | 7
  SBP, Standing 3 min, <90 mmHg | 3
  SBP, Standing 3 min, CFB ≥30 mmHg | 8
  SBP, Standing 3 min, CFB ≤ -30 mmHg | 4
  DBP, Supine, <50 mmHg | 2
  DBP, Supine, CFB ≥20 mmHg | 8
  DBP, Supine, CFB ≤ -20 mmHg | 7
  DBP, Standing 1 min, <50 mmHg | 3
  DBP, Standing 1 min, CFB ≥20 mmHg | 6
  DBP, Standing 1 min, CFB ≤ -20 mmHg | 7
  DBP, Standing 3 min, <50 mmHg | 2
  DBP, Standing 3 min, CFB ≥20 mmHg | 6
  DBP, Standing 3 min, CFB ≤ -20 mmHg | 6

3. Secondary Outcome: Number of Participants With PCS Electrocardiogram (ECG) Findings for QT Corrected According to Fridericia's Formula [QTcF])
Description: Number of participants with PCS postbaseline values for QTcF are categorized as follows: absolute value >450 milliseconds (msec) and ≤480msec; absolute value >480 msec and ≤500msec; absolute value >500 msec and increase from baseline >30 and ≤60 msec; increase from baseline >60 msec. Only those categories where at least 1 participant met the PCS criterion at least once during postbaseline are reported.
Time Frame: Up to 814 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SAGE-324
Number analyzed (Participants) | 97
Participants
  >450 msec and ≤480 msec | 9
  >480 msec and ≤500 msec | 3
  >500 msec | 1
  CFB >30 msec and ≤60 msec | 11
  CFB >60 msec | 2

4. Secondary Outcome: Number of Participants With PCS Laboratory Parameters
Description: Clinical laboratory test values are considered PCS if they meet either the lower-limit or higher-limit PCS criteria defined in the categories below. Number of participants with PCS laboratory values are summarized for clinical chemistry, liver function tests, hematology, and coagulation. Only those categories where at least 1 participant had a non-PCS value at Baseline and met the PCS criterion at least once during post-baseline are reported. Number analyzed is the number of participants with data available for analyses for the specified category.
Time Frame: Up to 814 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SAGE-324
Number analyzed (Participants) | 97
Participants
  Bicarbonate, Low: <18 millimoles per liter (mmol/L) | 1
  Calcium, High: >2.75 mmol/L | 1
  Glucose, Low: <2.8 mmol/L | 1
  Glucose, High: >13.9 mmol/L | 5
  Phosphate, Low: <0.61 mmol/L | 1
  Potassium, High: >5.4 mmol/L | 1
  Urea Nitrogen, High: >10.71 mmol/L | 11
  Alkaline Phosphatase, >1.5x Upper Limit of Normal (ULN) | 1
  Total Bilirubin, >1.5xULN | 2
  Total Bilirubin, >2xULN | 1
  Hematocrit, Low: <0.385 volume/volume (v/v) (Males): number analyzed (Participants) | 66
  Hematocrit, Low: <0.385 volume/volume (v/v) (Males) | 11
  Hematocrit, High: >0.55 v/v (Males): number analyzed (Participants) | 66
  Hematocrit, High: >0.55 v/v (Males) | 2
  Hematocrit, Low: <0.345 v/v (Females): number analyzed (Participants) | 31
  Hematocrit, Low: <0.345 v/v (Females) | 2
  Hemoglobin, Low: <115 grams/liter (g/L) (Males): number analyzed (Participants) | 66
  Hemoglobin, Low: <115 grams/liter (g/L) (Males) | 2
  Lymphocytes, Low: <0.5 10^9 cells per liter (10^9/L) | 2
  Neutrophils, Low: <1.5 10^9/L | 2
  Platelets, Low: <125 10^9/L | 2
  Activated Partial Thromboplastin Time (aPTT) (seconds), >1.5*ULN | 5
  Prothrombin Time (PT) (seconds), ≥1.11 x ULN | 18

5. Secondary Outcome: Change From Baseline in Epworth Sleepiness Scale (ESS) Score
Description: ESS consists of 8 items where participants rate, on a 4-point scale of 0 (no chance of dozing) to 3 (high chance of dozing), their usual chances of dozing off or falling asleep while engaged in 8 different activities. ESS total score is sum of the 8 individual item scores and estimates a participant's average sleep propensity. ESS score can range from 0 to 24. ESS score ≥ 10 was used to indicate excessive daytime sleepiness. A higher score indicates more severe excessive daytime sleepiness. Baseline was defined as last non-missing measurement prior to the first dose of investigational product. All participants received SAGE-324 according to a predefined up-titration scheme. Data was collected and reported in single arm for each participant who started treatment as specified and either completed or discontinued study.
Time Frame: Baseline, Days 8, 15, 22, 29, 36, 43, 50, 57, 70, 84, 112, 140, 168, 274, 365, 456, 548, 639, 730, 765, End of Treatment [EOT] (anytime, up to Day 793), End of Study [EOS] (anytime, up to Day 814)
Population: The Safety Set included all participants who were administered at least one dose of SAGE-324. Number analyzed is the number of participants with data available for analysis at specified timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAGE-324
Number analyzed (Participants) | 97
score on a scale
  Baseline | 5.0 (3.25)
  Change From Baseline at Day 8: number analyzed (Participants) | 94
  Change From Baseline at Day 8 | -0.4 (1.55)
  Change From Baseline at Day 15: number analyzed (Participants) | 95
  Change From Baseline at Day 15 | 0.0 (2.66)
  Change From Baseline at Day 22: number analyzed (Participants) | 94
  Change From Baseline at Day 22 | 0.2 (2.95)
  Change From Baseline at Day 29: number analyzed (Participants) | 95
  Change From Baseline at Day 29 | 0.3 (3.08)
  Change From Baseline at Day 36: number analyzed (Participants) | 89
  Change From Baseline at Day 36 | 1.0 (3.89)
  Change From Baseline at Day 43: number analyzed (Participants) | 87
  Change From Baseline at Day 43 | 0.9 (3.39)
  Change From Baseline at Day 50: number analyzed (Participants) | 87
  Change From Baseline at Day 50 | 1.0 (4.23)
  Change From Baseline at Day 57: number analyzed (Participants) | 80
  Change From Baseline at Day 57 | 0.7 (3.55)
  Change From Baseline at Day 70: number analyzed (Participants) | 76
  Change From Baseline at Day 70 | 0.7 (3.35)
  Change From Baseline at Day 84: number analyzed (Participants) | 71
  Change From Baseline at Day 84 | 0.8 (3.31)
  Change From Baseline at Day 112: number analyzed (Participants) | 67
  Change From Baseline at Day 112 | 0.3 (2.42)
  Change From Baseline at Day 140: number analyzed (Participants) | 54
  Change From Baseline at Day 140 | 0.0 (2.40)
  Change From Baseline at Day 168: number analyzed (Participants) | 50
  Change From Baseline at Day 168 | 0.3 (2.79)
  Change From Baseline at Day 274: number analyzed (Participants) | 40
  Change From Baseline at Day 274 | 0.4 (3.11)
  Change From Baseline at Day 365: number analyzed (Participants) | 25
  Change From Baseline at Day 365 | -0.5 (3.23)
  Change From Baseline at Day 456: number analyzed (Participants) | 16
  Change From Baseline at Day 456 | -0.1 (2.82)
  Change From Baseline at Day 548: number analyzed (Participants) | 7
  Change From Baseline at Day 548 | -1.3 (1.80)
  Change From Baseline at Day 639: number analyzed (Participants) | 6
  Change From Baseline at Day 639 | -1.5 (3.21)
  Change From Baseline at Day 730: number analyzed (Participants) | 3
  Change From Baseline at Day 730 | 1.7 (1.53)
  Change From Baseline at Day 765: number analyzed (Participants) | 3
  Change From Baseline at Day 765 | -1.3 (2.52)
  Change From Baseline at EOT (anytime, up to Day 793): number analyzed (Participants) | 12
  Change From Baseline at EOT (anytime, up to Day 793) | 1.3 (3.39)
  Change From Baseline at EOS (anytime, up to Day 814): number analyzed (Participants) | 29
  Change From Baseline at EOS (anytime, up to Day 814) | -0.2 (2.90)

6. Secondary Outcome: Number of Participants With Change From Baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) Responses
Description: C-SSRS scale consists of baseline evaluation that assesses lifetime experience of participant with suicidal ideation & behavior, & post-baseline evaluation that focuses on suicidality since last study visit. C-SSRS included 'yes'/'no' responses for assessment of suicidal ideation and behavior as well as numeric ratings for severity of ideation, if present (from 1-5, with 5 being most severe). Higher score indicated more severe symptoms. If any of assessments in suicidal behavior are 'Yes', category is considered as 'Suicidal behavior'. If any of assessments in suicidal ideation is 'Yes', but all assessments in suicidal behavior are 'No', category is considered as 'Suicidal ideation'. Baseline: any 'Yes' in any question in suicidal ideation/behavior prior to first dose of investigational product, excluding lifetime assessments. Data is reported for only those timepoints where participants had at least one 'yes' response to suicidal ideation or suicidal behavior except at Baseline.
Time Frame: Baseline up to Day 814
Population: The Safety Set. Number analyzed are number of participants with data available at specified timepoint. All participants received SAGE-324 according to a predefined up-titration scheme. Data was collected and reported in single arm for each participant who started treatment as specified and either completed or discontinued study.
Measure: Count of Participants; unit: Participants
Arm/Group | SAGE-324
Number analyzed (Participants) | 97
Participants
  Baseline: No Suicidal Ideation/Behavior | 97
  Baseline: Suicidal Ideation | 0
  Baseline: Suicidal Behavior | 0
  Day 70: number analyzed (Participants) | 76
  Day 70: No Suicidal Ideation/Behavior | 74
  Day 70: Suicidal Ideation | 1
  Day 70: Suicidal Behavior | 1
  Day 84: number analyzed (Participants) | 70
  Day 84: No Suicidal Ideation/Behavior | 69
  Day 84: Suicidal Ideation | 1
  Day 84: Suicidal Behavior | 0
  Day 112: number analyzed (Participants) | 65
  Day 112: No Suicidal Ideation/Behavior | 63
  Day 112: Suicidal Ideation | 2
  Day 112: Suicidal Behavior | 0

7. Secondary Outcome: Physician Withdrawal Checklist (PWC-20) Scale Total Score
Description: PWC is based on 35-item Penn Physician Withdrawal Checklist that was developed to measure benzodiazepine and benzodiazepine-like discontinuation symptoms. PWC-20 is a shorter version of Penn Physician Withdrawal Checklist and is made up of a list of 20 symptoms (e.g., loss of appetite, nausea-vomiting, diarrhea, anxiety-nervousness, irritability) that are rated on a scale of 0 (not present) to 3 (severe). Total scores can range from 0 to 60; higher scores indicating more severe symptoms. PWC-20 assessments were conducted at EOT and EOS to monitor for presence of potential withdrawal symptoms following discontinuation of IP. EOT was defined as first available assessment after last dose of study treatment and within 1 day of last dose of study treatment. All participants received SAGE-324 according to a predefined up-titration scheme. Data was collected and reported in single arm for each participant who started treatment as specified and either completed or discontinued study.
Time Frame: EOT (anytime, up to Day 793), EOS (anytime, up to Day 814)
Population: The Safety Set included all participants who were administered at least one dose of SAGE-324. Number analyzed are unique number of participants out of all the assessed participants with data available at the specified timepoint. Different participants may have contributed data for each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAGE-324
Number analyzed (Participants) | 97
score on a scale
  EOT (anytime, up to Day 793): number analyzed (Participants) | 33
  EOT (anytime, up to Day 793) | 6.5 (7.33)
  EOS (anytime, up to Day 814): number analyzed (Participants) | 82
  EOS (anytime, up to Day 814) | 5.0 (6.14)

ADVERSE EVENTS:
Time Frame: Up to 814 days
Description: The Safety Set: all participants who were administered at least one dose of SAGE-324. All participants received SAGE-324 according to a predefined up-titration scheme as follows: 15 mg from Day 1 to Day 14, followed by up-titration to 30 mg from Day 15 to Day 28, then to 45 mg from Day 29 to Day 42, and then 60 mg starting on Day 43. Data was collected and reported in single arm for each participant who started treatment as specified and either completed or discontinued study.
Arm/Group | SAGE-324
All-Cause Mortality (participants affected / at risk) | 0/97
Serious Adverse Events (participants affected / at risk) | 6/97
Other Adverse Events (participants affected / at risk) | 86/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SAGE-324 (N=97)
Aphasia (Nervous system disorders) | 1
COVID-19 (Infections and infestations) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SAGE-324 (N=97)
Somnolence (Nervous system disorders) | 49
Dizziness (Nervous system disorders) | 15
Balance disorder (Nervous system disorders) | 8
Cognitive disorder (Nervous system disorders) | 6
Tremor (Nervous system disorders) | 6
COVID-19 (Infections and infestations) | 10
Urinary tract infection (Infections and infestations) | 8
Upper respiratory tract infection (Infections and infestations) | 5
Depression (Psychiatric disorders) | 7
Insomnia (Psychiatric disorders) | 6
Abnormal dreams (Psychiatric disorders) | 5
Fatigue (General disorders) | 11
Feeling abnormal (General disorders) | 7
Fall (Injury, poisoning and procedural complications) | 7
Diarrhea (Gastrointestinal disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can either be a party and subject to the same restrictions as the institution, or if not a party, the restrictions are described on the face of the contract (i.e., PI is a contractor of the institution; PI is part of a larger group of study personnel; institution has contracted with or otherwise bound all study personnel under confidentiality obligations and requirements to vest intellectual property to the institution).

DOCUMENTS (2):
  • Study Protocol (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT05366751/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT05366751/SAP_001.pdf